CLINICAL TRIAL: NCT05831514
Title: Developing a Mobile Application for the Care of Children With Gastrostomy and The Effect of the Application on Gastrostomy Complications, Parental Care Burden, Self-Efficacy, and Anxiety Levels
Brief Title: Developing a Mobile Application for the Care of Children With Gastrostomy and The Effect of the Application on Gastrostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Yahya ERGEZEN, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KoçVakfıBursu; 2023.6 (Other Grant/Funding Number: Vehbi Koç Foundation Nursing Fund Project Support Program)
Record Dates: First submitted 2023-03-29; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Neuromuscular Diseases; Gastrointestinal Diseases
Keywords: Care burden; Parent education; Gastrostomy, Nursing; M-health application; Self-efficacy
MeSH Terms: conditions — Neuromuscular Diseases; Gastrointestinal Diseases; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: The research type is a pre-test-repeated post-test randomized controlled single blind study.
Who Masked: Participant
Masking Description: In the study, it will be ensured that the parents participating in the research do not know which group they are in. Therefore, one-way blinding will be applied in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Parents who meet the inclusion criteria will be informed about the study and invited to participate in the study. Verbal and written consent will be obtained from parents who meet the inclusion criteria and agree to participate in the study. In the pretest, the Complications Checklist, Zarit Caregiver Burden Scale, General Self-Efficacy Scale, State/Trait Anxiety Scale are completed by the parents. The mobile application will be introduced to the parents and they will be allowed to download it to their phones. Parents will be ensured to actively use the mobile application for three months. At the first month follow-up, the Complications Checklist, Zarit Caregiver Burden Scale, General Self-Efficacy Scale, State/Trait Anxiety Scale are completed by the parents. In the post-test, the Complications Checklist, Zarit Caregiver Burden Scale, General Self-Efficacy Scale, State/Trait Anxiety Scale are completed by the parents.
  Interventions: Other: Mobile Application Supported Education Program (G-MUEP)
- Control Group (No Intervention): Parents who meet the inclusion criteria will be informed about the study and invited to participate in the study. Verbal and written consent will be obtained from parents who meet the inclusion criteria and agree to participate in the study. In the pretest, the Complications Checklist, Zarit Caregiver Burden Scale, General Self-Efficacy Scale, State/Trait Anxiety Scale are completed by the parents. At the first month follow-up, the Complications Checklist, Zarit Caregiver Burden Scale, General Self-Efficacy Scale, State/Trait Anxiety Scale are completed by the parents. In the post-test, the Complications Checklist, Zarit Caregiver Burden Scale, General Self-Efficacy Scale, State/Trait Anxiety Scale are completed by the parents.

INTERVENTIONS:
Other: Mobile Application Supported Education Program (G-MUEP) — Parents who meet the inclusion criteria will use the Mobile Application Supported Education Program (G-MUEP).
  Arms: Intervention Group

SUMMARY:
Parents of children with gastrostomy have problems with the selection and preparation of nutritional products and catheter care during home care. Parents express that they want to receive practical training in the process of home care of the child with gastrostomy, they want to communicate more with the team and they need continuous monitoring to solve the problems encountered effectively. In this context, it is aimed to establish an appropriate training programme for the care of children with gastrostomy, to provide counselling and follow-up.

Digital health technologies are divided into different sub-branches. Mobile health applications constitute one of these structures. Mobile health applications are used in elective surgical interventions in pediatric surgery (tonsillectomy, hernia repair, circumcision, etc.) and in the home care process after organ transplantation. In pediatric surgery, many mobile health applications have been developed to support pain management, symptom monitoring, medication adherence, support care processes, postoperative follow-up and self-management processes. In mobile health applications, no mobile application has been found for the use of parents of children with gastrostomy. In Turkey, there is no known nursing study for the use of parents of children with gastrostomy. The aim of this study is to develop a mobile application for the care of children with gastrostomy and to determine the effect of the application on gastrostomy complications, care burden of parents, self-efficacy and anxiety level.

DETAILED DESCRIPTION:
Parents of children with gastrostomy have problems with the selection and preparation of nutritional products and catheter care during home care. Parents express that they want to receive practical training in the process of home care of the child with gastrostomy, they want to communicate more with the team and they need continuous monitoring to solve the problems encountered effectively. In this context, it is aimed to establish an appropriate training programme for the care of children with gastrostomy, to provide counselling and follow-up.

Digital health technologies are divided into different sub-branches. Mobile health applications constitute one of these structures. Mobile health applications are used in elective surgical interventions in pediatric surgery (tonsillectomy, hernia repair, circumcision, etc.) and in the home care process after organ transplantation. In pediatric surgery, many mobile health applications have been developed to support pain management, symptom monitoring, medication adherence, support care processes, postoperative follow-up and self-management processes. In mobile health applications, no mobile application has been found for the use of parents of children with gastrostomy. In Turkey, there is no known nursing study for the use of parents of children with gastrostomy. The aim of this study is to develop a mobile application for the care of children with gastrostomy and to determine the effect of the application on gastrostomy complications, care burden of parents, self-efficacy and anxiety level.

This research was planned in two stages as follows:

In the first stage, it was aimed to develop a mobile application supported education programme (G-MUEP) for the care of children with gastrostomy.

In the second stage, it was aimed to evaluate the effectiveness of G-MUEP.

For this purpose, the hypotheses of the research are as follows:

Parents using G-MUEP are more effective than the parents in the control group; Hypothesis 1 (H1): care burden is less. Hypothesis 2 (H1): their self-efficacy is higher. Hypothesis 3 (H1): anxiety levels are lower. Compared to the children in the control group, the children of the parents using G-MUEP; Hypothesis 1 (H1): gastrostomy-related complication findings are less.

ELIGIBILITY:
Inclusion Criteria:

* The gastrostomy was opened for the child within the last six months,
* The parent's willingness to participate in the study,
* The parent is literate in Turkish,
* Parental use of mobile devices,
* The parent has internet access,
* The parent has no communication barriers.

Exclusion Criteria:

-The parent has internet access problems.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-08-28 (Estimated)

PRIMARY OUTCOMES:
Complication Checklist | 3 Months
  A complication checklist consisting of 14 items was created by the researcher to determine the gastrostomy-related complications of the child with gastrostomy by reviewing the relevant literature.
Zarit Caregiver Burden Scale | 3 Months
  Zarit Caregiver Burden Scale was developed by Zarit, Reever and Bach Peterson in 1980. It is used to assess the distress experienced by caregivers of individuals in need of care. The scale is a Likert-type scale ranging from 1 to 5 as 'never', 'rarely', 'sometimes', 'often' or 'almost always'. Özlü, Yıldız & Aker (2009), who adapted the scale into Turkish, found the Cronbach's alpha coefficient of the scale to be 0.83 (Özlü, Yıldız, & Aker, 2009). A minimum score of zero and a maximum score of 76 can be obtained from the scale. The items in the scale are generally related to the social and emotional domain, and a high scale score indicates that the distress experienced is high.
General Self-Efficacy Scale | 3 Months
  The General Self-Efficacy Scale, developed by Schwarzer and Jarusalem in 1995 and validated by Aypay (2010) in Turkish, consists of 10 items in total. The scale, whose response category consists of a 4-point scale, is scored as "Completely wrong = 1 point", "Somewhat correct = 2 points", "Moderately correct = 3 points", and "Completely correct = 4 points". There are no reverse items and no cut-off points in the scale. The minimum score is 10 and the maximum score is 40. As the scale score increases, perceived self-efficacy increases. The Cronbach's alpha coefficient calculated in the Turkish validity-reliability study was found to be 0.83.
State/Trait Anxiety Scale | 3 Months
  State-Trait Anxiety Inventory will be used to measure the anxiety level of the parents. The State-Trait Anxiety Inventory was developed by Spielberger et al. (1970), translated into Turkish by Necla Öner and Le Compte in 1985, and its validity and reliability were tested in different groups. The scale can be applied to individuals over the age of 14. The State/Trait Anxiety Scale includes 40 statements that individuals can use to express their feelings. Depending on how the individual feels and the severity of his/her emotions, it is possible to rate them as "Not at all" (1), "A little" (2), "Quite a bit" (3), "Completely" (4) should mark one of the options.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Suluhan D, Yildiz D, Surer I, Fidanci Eren B, Balamtekin N. Effect of Gastrostomy Tube Feeding Education on Parents of Children with Gastrostomy. Nutr Clin Pract. 2021 Dec;36(6):1220-1229. doi: 10.1002/ncp.10586. Epub 2020 Oct 13. PMID 33047836
- [Background] Pars H, Cavusoglu H. A Literature Review of Percutaneous Endoscopic Gastrostomy: Dealing With Complications. Gastroenterol Nurs. 2019 Jul/Aug;42(4):351-359. doi: 10.1097/SGA.0000000000000320. PMID 29219857
- [Background] Kahveci G, Akin S. Knowledge Levels and Practices About the Enteral Nutritional Practices of Informal Caregivers Caring for Patients Fed Through a Percutaneous Endoscopic Gastrostomy Tube: A Descriptive Observational Study. Gastroenterol Nurs. 2021 Sep-Oct 01;44(5):E80-E90. doi: 10.1097/SGA.0000000000000623. PMID 34269704
- [Background] Fuchs S. Gastrostomy Tubes: Care and Feeding. Pediatr Emerg Care. 2017 Dec;33(12):787-791. doi: 10.1097/PEC.0000000000001332. PMID 29194216
- [Background] Bischoff SC, Austin P, Boeykens K, Chourdakis M, Cuerda C, Jonkers-Schuitema C, Lichota M, Nyulasi I, Schneider SM, Stanga Z, Pironi L. ESPEN practical guideline: Home enteral nutrition. Clin Nutr. 2022 Feb;41(2):468-488. doi: 10.1016/j.clnu.2021.10.018. Epub 2021 Nov 24. PMID 35007816
- [Background] Blumenstein I, Shastri YM, Stein J. Gastroenteric tube feeding: techniques, problems and solutions. World J Gastroenterol. 2014 Jul 14;20(26):8505-24. doi: 10.3748/wjg.v20.i26.8505. PMID 25024606
- [Background] Choi EK, Jung E, Ji Y, Bae E. A 2-Step Integrative Education Program and mHealth for Self-Management in Korean Children with Spina Bifida: Feasibility Study. J Pediatr Nurs. 2019 Nov-Dec;49:e54-e62. doi: 10.1016/j.pedn.2019.09.002. Epub 2019 Sep 10. PMID 31519400
- [Background] Pars H, Soyer T. Home Gastrostomy Feeding Education Program: Effects on the Caregiving Burden, Knowledge, and Anxiety Level of Mothers. JPEN J Parenter Enteral Nutr. 2020 Aug;44(6):1029-1037. doi: 10.1002/jpen.1747. Epub 2019 Nov 21. PMID 31755137